CLINICAL TRIAL: NCT05792410
Title: An Open, Multicenter Phase Ⅰb/Ⅱ Clinical Study of SHR-A1811 Combined With Dalpiciclib, Fulvestrant, Bevacizumab or Letrozole/Anastrozole in Patients With HER2 Low Advanced or Metastatic Breast Cancer.
Brief Title: A Phase Ⅰb/Ⅱ Clinical Study of SHR-A1811 Combined With Other Therapies in Patients With HER2 Low Advanced or Metastatic Breast Cancer.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-206
Record Dates: First submitted 2023-02-17; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-02

CONDITIONS: HER2 Low Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Bevacizumab

STUDY DESIGN:
Intervention Model Description: An open, multicenter, dose-finding and dose expansion investigational Phase IB/II clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-A1811 combined with Dalpiciclib Isethionate Tablets (Experimental)
  Interventions: Drug: SHR-A1811 & Dalpiciclib Isethionate Tablets
- SHR-A1811 combined with Fulvestrant (Experimental)
  Interventions: Drug: SHR-A1811 & Fulvestrant
- SHR-A1811 combined with Bevacizumab injection (Experimental)
  Interventions: Drug: SHR-A1811 & Bevacizumab injection

INTERVENTIONS:
Drug: SHR-A1811 & Dalpiciclib Isethionate Tablets — SHR-A1811：Lyophilized powder injection, 100mg / bottle, intravenous drip Dalpiciclib Isethionate Tablets：Tablet, 25mg / tablet, 50mg / tablet, 125mg / tablet, 150mg / tablet, oral
  Arms: SHR-A1811 combined with Dalpiciclib Isethionate Tablets
Drug: SHR-A1811 & Fulvestrant — SHR-A1811：Lyophilized powder injection, 100mg / bottle, intramuscular Fulvestrant：Injection, 5 ml: 0.25g/bottle, intramuscular
  Arms: SHR-A1811 combined with Fulvestrant
Drug: SHR-A1811 & Bevacizumab injection — SHR-A1811：Lyophilized powder injection, 100mg / bottle, intravenous drip Bevacizumab injection: injection, 100mg / bottle, intravenous drip
  Arms: SHR-A1811 combined with Bevacizumab injection

SUMMARY:
This study aims to evaluate the safety, tolerability, PK and preliminary anti-tumour activity of SHR-A1811 combined with other therapies in patients with HER2 low advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent, signed and dated IRB/EC approved informed consent, willing and able to comply with treatment planning visits, tests and other procedural requirements
2. When signing the informed consent, the age is 18-75 years old (including both ends), female patients who have pathologically documented HER2 low breast cancer
3. ECOG Performance Status of 0 or 1
4. Patient must have adequate tumor sample for biomarker assessment
5. At least one measurable lesion
6. Adequate organ function

Exclusion Criteria:

1. There are untreated or active central nervous system (CNS) tumor metastases
2. There was a third space effusion that could not be controlled by drainage (such as a large number of ascites, pleural effusion and pericardial effusion)
3. Major surgery within 4 weeks prior to enrollment
4. Has multiple primary malignancies within 5 years, excluding cured basal cell carcinoma of skin, cervical carcinoma in situ, papillary thyroid carcinoma, etc
5. Has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out at screening
6. Uncontrolled intercurrent illness
7. Uncontrolled or significant cardiovascular disease
8. Has known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection.
9. According to NCI-CTCAE v5.0 classification, those who have not recovered to grade Ⅰ toxicity caused by previous anti-tumour treatment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-02-27 (Estimated); Study Completion 2025-02-27 (Estimated)

PRIMARY OUTCOMES:
DLT(Phase I (dose-finding phase) main study endpoint) | At the end of cycle 1(each cycle is 28 days for SHR-A1811+ fulvestrant; each cycle is 21 days for SHR-A1811+other therapies.
AE(Phase I (dose-finding phase) main study endpoint) | Up to follow-up period, approximately 24 months
Incidence and severity of serious adverse events (SAE)(Phase I (dose-finding phase) main study endpoint) | Up to follow-up period, approximately 24 months
Objective response rate(The main end points of the second stage (efficacy expansion stage)) | Until progression, assessed up to approximately 24 months

SECONDARY OUTCOMES:
SHR-A1811 sparse PK concentrations in serum | While on study drug up to study completion, approximately 24 months
Dalpiciclib sparse PK concentrations in plasm | While on study drug up to study completion, approximately 24 months
Incidence of anti-drug antibodies (ADA) to SHR-A1811 over time | Up to follow-up period, approximately 24 months
Incidence of neutralizing antibody (NAb) to SHR-A1811 over time | Up to follow-up period, approximately 24 months
Duration of response (DoR) | Until progression or death, assessed up to approximately 24 months
Progression-free survival (PFS) | Until progression or death, assessed up to approximately 24 months

IPD SHARING:
Plan to Share IPD: Undecided